CLINICAL TRIAL: NCT01950416
Title: Pharmacodynamic Assessment of Ticagrelor vs High Dose Clopidogrel in Patients With ST Elevation Myocardial Infarction Exhibiting High Platelet Reactivity Post Fibrinolysis
Brief Title: Ticagrelor vs High Dose Clopidogrel in Patients With ST Elevation Myocardial Infarction Post Fibrinolysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-14
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: ST Elevation Myocardial Infarction; Fibrinolysis; P2Y12 Inhibitor
Keywords: ST elevation myocardial infarction; Fibrinolysis; Ticagrelor; Clopidogrel; Platelet reactivity
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 180mg loading dose (LD), followed by a 90mg x2 maintenance dose (MD) starting 12±6 hours post LD, until discharge.
  Interventions: Drug: Ticagrelor 180mg loading dose and 90mg bid maintenance dose
- Clopidogrel (Active Comparator): Clopidogrel 600mg loading dose (LD), followed by a 150mg once daily maintenance dose (MD) starting 12±6 hours post LD, until discharge.
  Interventions: Drug: Clopidogrel 600mg loading dose and 150mg maintenance dose

INTERVENTIONS:
Drug: Ticagrelor 180mg loading dose and 90mg bid maintenance dose
  Arms: Ticagrelor
Drug: Clopidogrel 600mg loading dose and 150mg maintenance dose
  Arms: Clopidogrel

SUMMARY:
This is a two-center, prospective, randomized, single-blind, investigator initiated, pharmacodynamic study of parallel design, carried out in 2 PCI-capable cardiology centers (Patras University Hospital and Konstantopoulio General Hospital of Athens).

Patients with ST elevation myocardial infarction, having undergone fibrinolysis in the previous 3 to 48 hours, who present high residual PR (defined as PRU ≥208 ) on admission, pre coronary angiography, will be randomized after written informed consent, in a 1:1 ratio to either:

Ticagrelor 180mg loading dose (LD), followed by a 90mg x2 maintenance dose (MD) starting 12±6 hours post LD, until discharge.

Or

Clopidogrel 600mg loading dose (LD), followed by a 150mg once daily maintenance dose (MD) starting 12±6 hours post LD, until discharge.

Platelet reactivity assessment will be performed at randomization (Hour 0) and at 2, 24 hours after randomization, as well as pre-discharge, using the VerifyNow assay, in platelet reactivity units (PRU).

Documentation of major adverse cardiac events (death, myocardial infarction, stroke, ischemia driven revascularization procedure with PCI or CABG) and bleeding (according to BARC criteria) will be performed until patient's discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old
2. Patients with STEMI, having undergone fibrinolytic therapy in the previous 3 to 48 hours
3. Presenting HPR (≥208 PRU) post 300mg clopidogrel loading dose ( assessment immediately before coronary angiography)
4. Informed consent obtained in writing

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Inability to give informed consent
* Cardiogenic shock
* Major periprocedural complications (death, stent thrombosis, vessel perforation, arrhythmias requiring cardioversion, temporary pacemaker insertion or intravenous antiarrhythmic agents, respiratory failure requiring intubation, vascular injury (arteriovenous shunt, retroperitoneal bleeding), major bleeding (need for bood transfusion or drop in haemoglobin post-PCI by ≥ 5 gr/ dl or intracranial bleeding)
* Known hypersensitivity to ticagrelor or clopidogrel
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 3 months.
* Other bleeding diathesis, or considered by investigator to be at high risk for bleeding
* Any previous history of stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
* Thombocytopenia (<100.000 / μL) at randomization
* Anaemia (Hct <30%) at randomization
* Polycytaemia (Hct > 52%) at randomization
* Periprocedural IIb/IIIa inhibitors administration
* Per os anticoagulants
* Recent (< 6 weeks) major surgery or trauma, including GABG.
* Subjects receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study.
* Concomitant oral or IV therapy with strong CY P3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazana vir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin /rifampicin, phenytoin, carbamazepine).
* Increased risk of bradycardiac events.
* Dialysis required.
* Severe uncontrolled chronic obstructive pulmonary disease
* Known severe hepatic impairement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity at 2 hours post randomization between the 2 treatment arms | 2 hours
  Platelet reactivity at 2 hours post randomization between the 2 treatment arms

SECONDARY OUTCOMES:
Platelet reactivity at 24 hours post randomization between the 2 treatment arms. | 24 hours
Platelet reactivity pre-discharge between the 2 treatment arms | 5 days
High on treatment platelet reactivity (HPR) rate (≥208 PRU) at 2 hours post randomization | 2 hours
High on treatment platelet reactivity (HPR) rate (≥208 PRU) at 24 hours post randomization | 24 hours
High on treatment platelet reactivity (HPR) rates (≥208 PRU) pre discharge | 5 days

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Konstantopoulio General Hospital of Athens, Athens, Attica
  - Patras University Hospital, Pátrai